CLINICAL TRIAL: NCT02766738
Title: Improving Mobility in Residential Aged Care: Comparing the Benefits of Two Resistance Exercise Programs
Brief Title: Improving Mobility in Residential Aged Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bond University (Other)
Responsible Party: Principal Investigator, Samantha Fien, PhD Student, Bond University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: RO1823
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Geriatric Disorder
Keywords: residential aged care; mobility; social participation; functional capability
MeSH Terms: interventions — Gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): All participants assigned to the control group will be given the option to engage in other activities that were offered by the facility during the 24-week intervention period. However, no specific resistance exercises were offered in these activities.
- GrACE program (Experimental): Participants in the exercise group will perform twice weekly training for 24 weeks. In brief, the program will include weight-bearing exercises and a range of seated, non-resisted upper- and lower-body dynamic and reaching movements. The following-weight bearing and resistance exercises: chair stands, chair dips, calf raises and hip flexor/abdominal lifts, trunk twists, and bicep curl and shoulder press. In total the sessions will be 45 minutes twice weekly.
  Interventions: Other: GrACE program
- GrACE + gait program (Experimental): GrACE program as mentioned above plus focus on gait specific training will be one-hour training sessions for 24 weeks. Gait exercises will be a combination of exercises: heel and toe raises, stepping in different directions, single leg stand¬ing, step-ups, and task-specific balance work (e.g. reaching outward from the base of support while standing, sitting, and standing and turning). Gait exercises will be upgraded by: 1) reducing hand support and/or 2) narrowing the base of support, and/or 3) introducing a cognitive challenge (e.g. counting backwards while performing exercise) or perform¬ing exercise with the eyes closed.
  Interventions: Other: GrACE + gait

INTERVENTIONS:
Other: GrACE program — to compare with the GrACE + gait programme in RAC, as well as the secondary objective of measuring the programme benefits on gait speed, sit to stand and handgrip strength against the intervention and control group
  Arms: GrACE program
Other: GrACE + gait — to compare with the GrACE programme in RAC, as well as the secondary objective of measuring the programme benefits on gait speed, sit to stand and handgrip strength against the intervention and control group
  Arms: GrACE + gait program

SUMMARY:
This study aims to test which of three exercise programs, previously demonstrated valuable for residential aged care adults, has the greatest benefit for walking speed and the spatiotemporal parameters that define it. The programs to be included are:

1. The GrACE program and
2. The GrACE plus Gait specific training.

DETAILED DESCRIPTION:
This study will employ a non-randomised controlled design in which three different 24-week exercise programs and a non-exercising control group will be compared in the residential aged care (RAC) setting. The three programs are the GrACE and the GrACE plus a gait specific training program.

Data Collection

~40 participants from two RAC facilities will be recruited into the study. This number of participants will provide 80% statistical power to identify moderate effect size between group differences on the primary outcome measures. The control group will be drawn from each of the RAC facility approached receiving exercise treatment. Participation will be informed by a discussion with the facilities Service Manager about the eligibility of participants and a medical history screen undertaken. All participants will provide informed written consent prior to participation.

Participants in the exercise group will perform twice weekly training for 24 weeks. Data will be collected at 0 weeks, 12 weeks and 24 weeks in the control and exercise groups.

ELIGIBILITY:
Inclusion Criteria:

* aged over 65 years
* residing in a RAC facility
* able to walk with a walker and/or walking stick or can self-ambulate for the test (including those who have had knee and hip replacements)
* can provide informed consent (Self- or by proxy).

Exclusion Criteria:

* end-stage terminal and/or life expectancy <6-months (ethical reasons)
* two person transfer or unable to self-ambulate (increased falls risk)
* unable to communicate or follow instructions (personal needs beyond the scope of this project)
* dangerous behaviours (endanger the client or research staff).

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Gait speed and spatio-temporal parameters (in a wider variety of walking tasks) | change from baseline to 24 weeks
  Gait speed and spatio-temporal parameters will be recorded via the GaitMat II system (Manufacturer is EQInc; Model is GaitMat II), which required participants to walk across a level pressure mat system 3.66 m (11.91 ft.) long (McDonough et al. 2001). Participants completed the trials at their preferred (habitual) walking (gait) speed. All measures will be initiated from a standing start 2 m (6.56 ft.) from the GaitMat II platform as suggested by Kressig and Beauchet (Kressig & Beauchet 2006) to reduce the effect that acceleration may have on gait speed. Three conditions will be measured which include normal walking, along with two dual tasks. These dual tasks include: (i) walking while carrying a glass of water in the participants preferred hand, (ii) walking while counting backwards from 30. Each of these gait conditions will be performed for three repetitions in a randomised block order (Taylor, 2012).

SECONDARY OUTCOMES:
Sit to stand performance | change from baseline to 24 weeks
  In the sit-to-stand measure, participants sat and stood to a full standing position from a chair as many times as possible in 30 seconds whilst keeping their arms crossed against their chest (Millor 2013). Measurement units = repetitions in 30 seconds
handgrip strength | change from baseline to 24 weeks
  Upper body muscle function was measured by isometric handgrip strength and sit-to-stand performance, respectively. When performing the handgrip strength assessments, participants were seated, instructed to keep their elbow at 90° and asked to squeeze a handgrip dynamometer (Sammons Preston Roylan, Bolingbrook, IL) to their maximum ability for a period of up to five seconds (Mathiowetz 2002). Three trials were performed with the subject's dominant hand with one-minute rest between trials and the best result used for analysis (Roberts 2011). Measurement units = kilograms
Body Composition | change from baseline to 24 weeks
  measure the volume of lean body mass (kg) and fat mass (kg) and the skeletal muscle index will be calculated using the BIA.
Quality of Life (EQ-5D-EL) | change from baseline to 24 weeks
  The EQ-5D-EL descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels: no problems, some problems and extreme problems.
Sarcopenia status (SARC-F) | change from baseline to 24 weeks
  The SARC-F questionnaire is a rapid diagnostic test used to screen individuals for sarcopenia. There are five SARC components: strength, assistance with walking, rising from a chair, climbing stairs, and falls. The scores range from 0 to 2 points for each of the five components, allowing a total score of 0-10. Studies have suggested that a score equal to or greater than four is predictive of sarcopenia and poor health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Keogh, PhD, Principal Investigator — Bond University
Locations (1):
- Darlington RSL Care, Tweed Heads, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mathiowetz V. Comparison of Rolyan and Jamar dynamometers for measuring grip strength. Occup Ther Int. 2002;9(3):201-9. doi: 10.1002/oti.165. PMID 12374997
- [Result] McDonough AL, Batavia M, Chen FC, Kwon S, Ziai J. The validity and reliability of the GAITRite system's measurements: A preliminary evaluation. Arch Phys Med Rehabil. 2001 Mar;82(3):419-25. doi: 10.1053/apmr.2001.19778. PMID 11245768
- [Result] Kressig RW, Beauchet O; European GAITRite Network Group. Guidelines for clinical applications of spatio-temporal gait analysis in older adults. Aging Clin Exp Res. 2006 Apr;18(2):174-6. doi: 10.1007/BF03327437. PMID 16702791
- [Result] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Result] Millor N, Lecumberri P, Gomez M, Martinez-Ramirez A, Izquierdo M. An evaluation of the 30-s chair stand test in older adults: frailty detection based on kinematic parameters from a single inertial unit. J Neuroeng Rehabil. 2013 Aug 1;10:86. doi: 10.1186/1743-0003-10-86. PMID 24059755
- [Result] Taylor ME, Delbaere K, Mikolaizak AS, Lord SR, Close JC. Gait parameter risk factors for falls under simple and dual task conditions in cognitively impaired older people. Gait Posture. 2013 Jan;37(1):126-30. doi: 10.1016/j.gaitpost.2012.06.024. Epub 2012 Jul 23. PMID 22832468
- [Result] Hewitt J, Refshauge KM, Goodall S, Henwood T, Clemson L. Does progressive resistance and balance exercise reduce falls in residential aged care? Randomized controlled trial protocol for the SUNBEAM program. Clin Interv Aging. 2014 Feb 21;9:369-76. doi: 10.2147/CIA.S53931. eCollection 2014. PMID 24591821